CLINICAL TRIAL: NCT04204993
Title: Assessment of Wearable Sensors During Experimental Human Influenza Infection (Sigma Plus)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Duke University (Other); RTI International (Other); Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19HH5451
Record Dates: First submitted 2019-11-12; First posted 2019-12-19 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Influenza A H3N2
Keywords: Influenza A H3N2

STUDY DESIGN:
Intervention Model Description: Biological: Influenza A/Belgium/4217/2015 at a dose of 5x105 TCID50 in a volume of 0.5 milliliters via intranasal drops
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental: Influenza A (Experimental): Participants will be inoculated with Influenza A/Belgium/4217/2015 at a dose of 5x105 TCID50 in a volume of 0,5mL via intranasal drops or spray. They will then be monitored as in-patients for 10 days with daily clinical assessment and blood, respiratory tract sampling, and sensor monitoring. Following discharge, they will be followed up for up to 6 months post-inoculation.
  Interventions: Device: Lumee Oxygen Platform

INTERVENTIONS:
Device: Lumee Oxygen Platform — Two sensors will be inserted (one in the skin fo the upper arm and one on the side of the chest). A wireless patch reader is placed on top of the skin over the area where the sensor has been placed to measure local oxygen content.

SUMMARY:
The aim of the study is to investigate disease in volunteers deliberately infected with influenza A(H3N2), including biological markers of inflammation and immune response, and changes in physiological parameters including heart rate, respiratory rate, physical activity, oxygen saturation and electrocardiographic data during the onset of influenza infection. Ultimately, this may lead to prediction of symptomatic disease at an earlier stage to allow more effective interventions. The experimental medicine study design will involve human influenza infection challenge, whereby volunteers will be inoculated with influenza virus and monitored in hospital for 10 days as they develop and get better from flu. Continuously-monitoring wearable physiological sensors will be given to the participants 7 days before this and worn continuously until the end of the flu infection.

DETAILED DESCRIPTION:
Influenza ('flu') is one of the most common causes of severe lung infection. Seasonal flu affects between 10 and 46% of the population each year and causes around 12 deaths in every 100,000 people infected. Furthermore, new strains of flu viruses emerge unpredictably every few years, causing pandemics that spread rapidly across the world. Since currently available antiviral drugs and vaccines cannot prevent these outbreaks, it is essential to be able to identify flu infections at an early stage to enable rapid treatment of individuals and implementation of public health measures.

The aim of the study is to investigate disease in volunteers deliberately infected with influenza A(H3N2), including biological markers of inflammation and immune response, and changes in physiological parameters including heart rate, respiratory rate, physical activity, oxygen saturation and electrocardiographic data during the onset of influenza infection. To achieve this, the investigators will recruit healthy volunteers and inoculate them with a flu virus, after which they will be observed in hospital while they develop a cold. Each volunteer will be given a number of devices that they will wear before and during infection. In addition, they will have blood and nasal samples taken to examine the way their immune system responds to infection. The resulting data will be analysed to see if the sensors data correlate with the onset of infection and these will be compared with measures of the immune response. Ultimately, the investigators anticipate that optimised sensor data from devices to be developed may be useful in rapidly detecting when someone is about to develop flu infection, so that they can quickly be treated and outbreaks may be identified at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons aged 18 to 55 years, able to give informed consent

Exclusion Criteria:

* Chronic respiratory disease (asthma, chronic obstructive pulmonary disease, rhinitis, sinusitis) in adulthood
* Inhaled bronchodilator or steroid use within the last 12 months
* Use of any medication or other product (prescription or over-the-counter) for symptoms of rhinitis or nasal congestion within the last 3 months
* Acute upper respiratory infection (URI or sinusitis) in the past 6 weeks
* Smoking in the past 6 months OR >5 pack-year lifetime history
* Subjects with allergic symptoms present at baseline
* Clinically relevant abnormality on chest X-ray
* Any ECG abnormality deemed clinically significant.
* Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 3 years, the elderly (>65 years), immunosuppressed persons, or those with chronic respiratory disease
* Subjects with known or suspected immune deficiency
* Receipt of systemic glucocorticoids (in a dose ≥ 5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within 6 months prior to challenge
* Known immunoglobulin A deficiency, immotile cilia syndrome, or Kartagener's syndrome
* History of frequent nose bleeds
* Any significant medical condition or prescribed drug deemed by the study doctor to make the participant unsuitable for the study
* Pregnant or breastfeeding women
* Positive urine drug screen
* Detectable baseline antibody titres against influenza challenge strains
* History of hypersensitivity to eggs, egg proteins, gentamicin, gelatin or arginine, or with life-threatening reactions to previous influenza vaccinations.
* Participants may only recruited if they have previously been involved in research if they have completed the earlier study and are beyond the washout period of any administered drugs or period of effect of any intervention that would cause interference for either study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with Duke university, and RTI International, such as ethnicity and age. It will be identifiable only by their unique study code, with no personal details.
Supporting Information: Study Protocol, CSR
Access Criteria: According to study protocol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 healthy volunteers were enrolled in the study and followed up from the period 11th February 2020 to 17th May 2021. The study was suspended from March to August 2020 due to the global SARS-CoV-2 pandemic.
Groups:
- Experimental: Influenza A: Participants were inoculated with Influenza A/Belgium/4217/2015 at a dose of 5x10^5 TCID50 in a volume of 0,5mL via intranasal drops. They were monitored as in-patients for 10 days with daily clinical assessment and blood, respiratory tract sampling, and sensor monitoring. Following discharge, they were followed up for 6 months post-inoculation.
  Lumee Oxygen Platform: Two sensors were inserted (one in the skin of the upper arm and one on the side of the chest). A wireless patch reader was placed on top of the skin over the area where the sensor was placed to measure local oxygen content.
Period: Overall Study
Arm/Group | Experimental: Influenza A
Started | 20
Group A | 4
Group B | 6
Group C | 6
Group D | 4
Completed | 20 (Last follow-up visit on Day 180.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Other than the 20 enrolled participants, there were some screening failures due to abnormal blood results, spirometry and chest x-ray.
Groups:
- Experimental: Influenza A: Participants were inoculated with Influenza A/Belgium/4217/2015 at a dose of 5x10^5 TCID50 in a volume of 0,5mL via intranasal drops. They were then monitored as in-patients for 10 days with daily clinical assessment and blood, respiratory tract sampling, and sensor monitoring. Following discharge, they were followed up for up to 6 months post-inoculation.
  Lumee Oxygen Platform: Two sensors were inserted (one in the skin for the upper arm and one on the side of the chest). A wireless patch reader was placed on top of the skin over the area where the sensor was placed to measure local oxygen content.
Arm/Group | Experimental: Influenza A
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White British | 7
  Ethnicity: White Irish | 2
  Ethnicity: White (all other) | 4
  Ethnicity: Black or Black British (African) | 1
  Ethnicity: Black or Black British (all other) | 1
  Ethnicity: Asian or Asian British (Indian) | 2
  Ethnicity: Asian or Asian British (Pakistani) | 1
  Ethnicity: Chinese | 1
  Ethnicity: All other ethnic groups | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of PCR-confirmed Influenza Infections
Description: Nasal wash viral load by quantitative polymerase chain reaction (qPCR)
Time Frame: Baseline to day 28
Population: One participant who was PCR positive for the challenge agent also tested positive for Rhinovirus on Day 4 post-inoculation therefore this participant was excluded from all further analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Influenza A: Participants were inoculated with Influenza A/Belgium/4217/2015 at a dose of 5x10^5 TCID50 in a volume of 0,5mL via intranasal drops. They were then monitored as in-patients for 10 days with daily clinical assessment and blood, respiratory tract sampling, and sensor monitoring. Following discharge, they were followed up for up to 6 months post-inoculation.
  Lumee Oxygen Platform: Two sensors were inserted (one in the skin fo the upper arm and one on the side of the chest). A wireless patch reader was placed on top of the skin over the area where the sensor was placed to measure local oxygen content.
Arm/Group | Experimental: Influenza A
Number analyzed (Participants) | 20
Participants
  PCR positive Influenza infection | 17
  PCR negative Influenza infection | 3

2. Secondary Outcome: Time to Algorithmic Detection of Heart Rate Abnormalities
Description: Sensor data read-outs
Time Frame: Baseline to day 10
Population: All metrics were expressed as z-scores matched for physical activity level. Multivariate process control techniques were used to quantify the change in the multidimensional HRV parameter space relative to baseline and formulated an algorithm for the detection of the illness. 170 total days monitored. Mean parameter values were computed on 24hr increments.
Measure: Mean (Standard Deviation); unit: hours post-inoculation
Groups:
- Experimental: Influenza A: Participants were inoculated with Influenza A/Belgium/4217/2015 at a dose of 5x10^5 TCID50 in a volume of 0,5mL via intranasal drops. They were then monitored as in-patients for 10 days with daily clinical assessment and blood, respiratory tract sampling, and sensor monitoring. Following discharge, they were followed up for up to 6 months post-inoculation.
  Lumee Oxygen Platform: Two sensors were inserted (one in the skin fo the upper arm and one on the side of the chest). A wireless patch reader was placed on top of the skin over the area where the sensor had been placed to measure local oxygen content.
Arm/Group | Experimental: Influenza A
Number analyzed (Participants) | 20
hours post-inoculation | 52 (17)

3. Secondary Outcome: Tissue Oxygen Levels
Description: Sensor data read-outs
Time Frame: Baseline to day 10
Population: Data collected with the Lumee devices per group (A, B, and D). Lumee devices were not used in Group C. LOI = Lumee Oxygen Index which is a measure proportional to micro-molar concentration of Oxygen in the interstitial fluid. The normal range for LOI is 10-52. A higher LOI corresponds to higher micro-molar concentration of Oxygen in the interstitial fluid.
Measure: Mean (Standard Deviation); unit: LOI
Groups:
- Group A: Participants were inoculated with Influenza A/Belgium/4217/2015 at a dose of 5x10^5 TCID50 in a volume of 0,5mL via intranasal drops. They were then monitored as in-patients for 10 days with daily clinical assessment and blood, respiratory tract sampling, and sensor monitoring. Following discharge, they were followed up for up to 6 months post-inoculation.
  Lumee Oxygen Platform: Two sensors were inserted (one in the skin fo the upper arm and one on the side of the chest). A wireless patch reader was placed on top of the skin over the area where the sensor was placed to measure local oxygen content.
- Group B; Group D: Participants were inoculated with Influenza A/Belgium/4217/2015 at a dose of 5x10^5 TCID50 in a volume of 0,5mL via intranasal drops. They were then monitored as in-patients for 10 days with daily clinical assessment and blood, respiratory tract sampling, and sensor monitoring. Following discharge, they were followed up for up to 6 months post-inoculation.
Arm/Group | Group A | Group B | Group D
Number analyzed (Participants) | 4 | 6 | 4
LOI | 12.6 (8.8) | 13.7 (8.5) | 12.5 (6.8)

4. Secondary Outcome: Participant-reported Total Symptom Score
Description: Cumulative daily symptom score derived from self-reported upper and lower respiratory and systemic symptoms by diary card using the modified Jackson's symptom scoring system. Eight symptoms were scored: nasal obstruction, nasal discharge, sore throat, sneezing, cough, malaise, headache, and chills. Each symptom was scored 0-3, where 0=absent, 1=mild, 2=moderate and 3=severe. The maximum daily score is 24 and minimum daily score is 0.
Time Frame: Day 1, Day 3 and Day 10
Population: 13 of 16 PCR positive participants (1 participant was excluded from the analysis due to co-infection with Rhinovirus) developed influenza-like symptom following inoculation. The 3 remaining participants were asymptomatic with modified Jackson's symptom scoring system.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Experimental: Influenza A
Number analyzed (Participants) | 19
scores on a scale
  Day 1 | 2.44 (2.76)
  Day 3 (peak) | 11.50 (13.67)
  Day 10 | 1.19 (2.69)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the study period, until the 6 month follow-up visit.
Description: Adverse event data was collected by observations and reports from study participants.
Groups:
- Experimental: Influenza A: Participants were inoculated with Influenza A/Belgium/4217/2015 at a dose of 5x10^5 TCID50 in a volume of 0,5mL via intranasal drops. They were then monitored as in-patients for 10 days with daily clinical assessment and blood, respiratory tract sampling, and sensor monitoring. Following discharge, they were followed up for up to 6 months post-inoculation.
  Lumee Oxygen Platform: Two sensors were inserted (one in the skin of the upper arm and one on the side of the chest). A wireless patch reader was placed on top of the skin over the area where the sensor was placed to measure local oxygen content.
Arm/Group | Experimental: Influenza A
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 9/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Influenza A (N=20)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Erythema caused ny patches noted on Lumee sites on lower right arm and upper left chest. Resolved spontaneously.
Dental issue (General disorders) | 1 (1) — Tooth cracked whilst eating. Visited dentist for dental treatment when symptoms were reduced and volunteer was past peak of infectious stage.
Foot injury (Skin and subcutaneous tissue disorders) | 1 (1) — Slipper caused old surgical wound on foot to blister and got infected. Swelling and erythema noticed on foot. Doctor prescribed oral antibiotic treatment. Problem resolved.
COVID symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Participant attended Day 28 treatment with recent symptoms of temperature, lethargy and cough. Participant was advised to return home to isolate and get tested for COVID-19. No samples were taken, Day 28 visit was delayed.
Cystoscopy (Renal and urinary disorders) | 1 (1) — Underwent cystoscopy December 2020 to investigate haematuria, with onset prior to the study. No abnormality detected and no further investigations required.
Rhinovirus positive (Infections and infestations) | 1 (1) — Tested positive for Rhinovirus on Day -1. Results not back in time for inoculation, so was inoculated with Influenza H3N2 on Day 0. Isolated in side room when results came back. Sampling and other tests were taken as per study protocol.
COVID-19 infection (Infections and infestations) | 2 (2) — Tested positive for COVID-19 during the global pandemic. Symptoms resolved within a couple of weeks without any need of healthcare support.
Ear infection (Infections and infestations) | 1 (1) — Earache on Day 180 follow-up visit. Clinically stable. Swelling and erythema with yellow discharge seen in ear on examination. Recommended to contact GP for further advise.

LIMITATIONS AND CAVEATS:
Lumee oxygen devices failed to charge on the charging stations provided. Advice and support were given by the engineering team but unable to resolve. No Lumee devices were used for participants SPFC011-SPFC016. The devices were shipped to manufacturer for further troubleshooting and investigation. The batteries were repaired, and the devices were returned to ICL for the remaining participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04204993/Prot_SAP_000.pdf